CLINICAL TRIAL: NCT02418702
Title: A Randomized Controlled Trial to Decrease Suicidal Thinking Using Ketamine
Brief Title: A Study to Decrease Suicidal Thinking Using Ketamine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI no longer at facility.
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMCSD.2014.0031
Record Dates: First submitted 2015-04-07; First posted 2015-04-16 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Depression; Suicide
Keywords: depression; suicide; ketamine; rapid intravenous bolus; sub-anesthetic dose; double-blind placebo control
MeSH Terms: conditions — Depression; Suicide | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.2mg/kg ketamine (Experimental): After being assessed, and giving informed consent, participants would receive 0.2mg/kg ketamine. Their suicidal thinking, depression, and other symptoms would be monitored acutely for 240 min after drug infusion, and the for lasting changes the next day, at hospital discharge, 2 weeks, and 10 weeks.
  Interventions: Drug: 0.2 mg/kg ketamine
- placebo (Placebo Comparator): After being assessed, and giving informed consent, participants would receive a placebo. Symptoms will be monitored.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: 0.2 mg/kg ketamine — 20 patients will randomly be assigned 0.2 mg/kg of Ketamine
  Other Names: Ketamine
  Arms: 0.2mg/kg ketamine
Other: placebo — 20 patients will randomly be assigned a placebo
  Arms: placebo

SUMMARY:
Depression treatment typically is slow acting. Patients presenting with acute suicidality have few immediate treatment options. However, sub-anesthetic doses of ketamine have been now widely tested as a rapid-acting treatment for depression. Gregory Larkin et al at Yale showed this could be applied to suicidal patients, with 14 of 15 participants showing remission of suicidal thinking within 40 min of the administration of ketamine, with 13 showing lasting remission out to 10 days. No serious side effects were reported. This project proposes to conduct a randomized, placebo-controlled trial of this, same intervention in military patients recently hospitalized for suicidal thinking. After being assessed, and giving informed consent, participants would receive 0.2mg/kg ketamine or placebo. Their suicidal thinking, depression, and other symptoms would be monitored acutely for 240 min after drug infusion, and the for lasting changes the next day, at hospital discharge, 2 weeks, and 10 weeks. Potential adverse events will be monitored via the electronic medical record for up to a year.

DETAILED DESCRIPTION:
Patients presenting for acute suicidality have few immediate treatment options to alleviate their suffering aside from psychiatric hospitalization for safety assurance. Therapy and psychiatry medication may decrease depression over time, but this does little to improve depression and suicidal thinking in the short term. Preliminary data from a recent study by Larkin et al at Yale University showed evidence to support a promising novel treatment modality with rapid effects on suicidal ideation for up to 10 days post infusion through the use of a single sub-anesthetic rapid intravenous bolus dose of ketamine (0.2-mg/kg) administered in the acute Emergency Department setting. This study showed favorable evidence to support further investigation into the use of a single sub-anesthetic bolus dose of ketamine in acutely depressed and/or suicidal patients in the emergency room setting. Based on the success of this study, Naval Medical Center San Diego (NMCSD) started the previously mentioned, small, unfunded randomized, placebo-controlled trial of this ketamine protocol for patients who were pending psychiatric hospitalization because of suicidal thinking. Data collection was highly flawed, but unpublished, preliminary results show that the ketamine treatment resulted in significant decreased in suicidal thinking.

Of note, there were no adverse events associated with the ketamine administration. Although the infusion was done in an Emergency Department (ED) setting, the patients were seated in clinic chairs, and required no additional monitoring or intervention beyond what could be provided in any clinic our psychiatric hospital setting. It is the intent of the project to expand on our unfunded trial, allowing us to treat a wider range of participants who come in to the psychiatric ward because of suicidal thinking. This study is being pursued in the context that existing therapies for major depression have a lag of onset of action of several weeks, resulting in an increased risk of possible and considerable morbidity and possibly mortality through suicide. This study would explore the efficacy of Ketamine's (a N-Methyl-D-aspartate (NMDA) receptor antagonist) rapid and potentially long-lasting antidepressant effects in a suicidal population. The Investigators hope to gather data that could potentially impact treatment practices in the military setting for acutely depressed patients. This may potentially shorten, delay, or even forgo admissions to the psychiatric ward in the future, as well as potentially reducing the long term suicidality.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily, psychiatrically hospitalized at NMCSD within the last 12 hours for suicidal thinking
* BSS greater than 4
* BHS greater than 8
* BDI greater than 19
* Ability to give informed consent
* Active duty military status
* Verified negative pregnancy test for females

Exclusion Criteria:

* Psychosis or bipolar disorder
* Pregnancy
* Involuntary status on presentation to the ED
* Positive for illicit drugs of abuse
* Blood alcohol level greater than zero
* Previous enrollees in this treatment protocol will be excluded from repeat participation
* Any patient brought for command directed psychiatric evaluation
* Specific contraindication to the use of ketamine are as follows and under such circumstances or conditions, personnel with the following should be excluded from participation in this study:

A) patients with elevated intracranial pressure, uncontrolled hypertension, coronary artery disease, aneurysms, thyrotoxicosis, congestive heart failure (CHF), a recent history of head or eye injury, or angina B) all personnel in whom a significant elevation of blood pressure would constitute a serious hazard to their overall health and well-being C) patients currently utilizing the following medications: conivaptan, dasatinib, peginterferon alfa-2b, quazepam, tocilizumab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Estimated); Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in baseline in depressive symptoms measured by Beck Scale for Suicide ideation (BSS), Beck Hopelessness Scale (BHS), and Beck Depression Index (BDI) | baseline and 240 minutes
  measure whether a significant reduction in depressive symptoms, as assessed by the BSS, BHS, and BDI occurs shortly after administration of ketamine
Change in baseline in depressive symptoms measured by Beck Scale for Suicide ideation (BSS), Beck Hopelessness Scale (BHS), and Beck Depression Index (BDI) | baseline and 2 weeks
Change in baseline in depressive symptoms measured by Beck Scale for Suicide ideation (BSS), Beck Hopelessness Scale (BHS), and Beck Depression Index (BDI) | baseline and 10 weeks

SECONDARY OUTCOMES:
Reduction in suicidal thinking measured by BSS, BHS, and BDI | 1 day post-infusion
  single bolus of ketamine's effect on sustained reduction of symptoms
Reduction in suicidal thinking measured by BSS, BHS, and BDI | 2 weeks post-infusion
Reduction in suicidal thinking measured by BSS, BHS, and BDI | 10 weeks post-infusion

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Capobianco, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

REFERENCES:
- [Background] Melville NA. Bolus dose of ketamine offers fast-acting alleviation of acute depression in ED setting. Medscape Medical News. September 29, 2010.
- [Background] Messer MM, Haller IV. Maintenance ketamine treatment produces long-term recovery from depression. Primary Psychiatry. 2010; 17(4):48-50.
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Yilmaz A, Schulz D, Aksoy A, Canbeyli R. Prolonged effect of an anesthetic dose of ketamine on behavioral despair. Pharmacol Biochem Behav. 2002 Jan-Feb;71(1-2):341-4. doi: 10.1016/s0091-3057(01)00693-1. PMID 11812542
- [Background] Sanacora G, Gueorguieva R, Epperson CN, Wu YT, Appel M, Rothman DL, Krystal JH, Mason GF. Subtype-specific alterations of gamma-aminobutyric acid and glutamate in patients with major depression. Arch Gen Psychiatry. 2004 Jul;61(7):705-13. doi: 10.1001/archpsyc.61.7.705. PMID 15237082
- [Background] Zarate CA Jr, Du J, Quiroz J, Gray NA, Denicoff KD, Singh J, Charney DS, Manji HK. Regulation of cellular plasticity cascades in the pathophysiology and treatment of mood disorders: role of the glutamatergic system. Ann N Y Acad Sci. 2003 Nov;1003:273-91. doi: 10.1196/annals.1300.017. PMID 14684452
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Panzer O, Moitra V, Sladen RN. Pharmacology of sedative-analgesic agents: dexmedetomidine, remifentanil, ketamine, volatile anesthetics, and the role of peripheral mu antagonists. Crit Care Clin. 2009 Jul;25(3):451-69, vii. doi: 10.1016/j.ccc.2009.04.004. PMID 19576524